CLINICAL TRIAL: NCT01767506
Title: A Surveillance and Azithromycin Treatment for Newcomers and Travelers Evaluation: The ASANTE Trial
Acronym: ASANTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00076305; U10EY022584 (NIH)
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Trachoma
Keywords: Trachoma; Azithromycin; Mass treatment
MeSH Terms: conditions — Trachoma | interventions — Therapeutics; Azithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Communities will receive usual care, including annual mass drug administration with azithromycin if trachoma infection level is greater than 1% or TF is 5% or more. Communities will have MDA stopped if infection is 1% or less, or TF is less than 5%. MDA will be reinstated if infection re-emerges to 6% or more. In addition, surveillance and treatment with azithromycin of newcomer and traveler families within 2 weeks of arrival to or return to the community.
  Interventions: Other: Surveillance and treatment with azithromycin of newcomer and traveler families; Other: Usual care
- Usual Care (Active Comparator): Communities will receive usual care, including annual mass drug administration with azithromycin if trachoma infection level is greater than 1% or TF is 5% or more. Communities will have MDA stopped if infection is 1% or less, or TF is less than 5%. MDA will be reinstated if infection re-emerges to 6% or more.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Surveillance and treatment with azithromycin of newcomer and traveler families — The intervention is a surveillance for newcomers and travelers in communities, and provision of azithromycin to them at the time of arrival, in advance of scheduled mass drug administration
  Other Names: Zithromax
  Arms: Intervention
Other: Usual care — Scheduled mass drug administration (MDA) of azithromycin if trachoma infection level is greater than 1% or TF is 5% or more. Communities will have MDA stopped if infection is 1% or less, or TF is less than 5%. MDA will be reinstated if infection re-emerges to 6% or more.
  Other Names: Zithromax

SUMMARY:
Infection with C. Trachomatis has decreased substantially in trachoma endemic areas following repeated annual mass drug administration (MDA) with azithromycin, although not as rapidly as anticipated. The investigators propose to conduct a clinical trial in 52 communities in Kongwa, Tanzania that on average have trachoma infection at 3.5%. The investigators plan that all communities would have annual rounds of MDA if infection is greater than 1% or follicular trachoma (TF) is 5% or more, but half would be randomized to a surveillance and treatment program to identify and treat new families and families who travel after mass treatment. Communities will have MDA stopped if infection is 1% or less, or TF is less than 5%. MDA will be reinstated if infection re-emerges to 6% or more. The proportion of communities that are able to stop mass treatment will be compared in the group of communities randomized to mass treatment plus the newcomer/traveler treatment program compared to the communities randomized to mass treatment alone after 24 months.

At the recommendation of the Data Safety and Monitoring Committee in March 2015, thirty eight (38) of the 52 communities identified as being at risk of trachoma re-emergence at 18 months will be surveyed at 30 months. At risk of trachoma re-infection communities have C. trachomatis infection rates less than or equal to 1% or TF < 5% at the time of the 18 month survey. Surveillance of communities for families that meet the newcomer or traveler status will extend 6 months beyond the 24 month survey to 30 months in the intervention communities only. A survey of sentinel children in the intervention and control communities at 30 months will be conducted to assess the level of trachoma and infection in all 38 communities at risk of trachoma re-emergence.

ELIGIBILITY:
Inclusion Criteria:

Census and Mass Drug Administration (MDA): All persons residing in the 52 study communities will be eligible for both the census and the annual mass azithromycin administrations.

Intervention: In the 26 intervention communities, active surveillance for new families and returning travelers will be undertaken, and those meeting the criteria below will be eligible for family treatment with azithromycin if:

Families are "newcomers" and

* They have children under 10 years of age
* They have moved into a new house in the community or into an existing household
* They plan to reside for at least 1 month in the study community and
* They have moved from a community that has not had an MDA in the last year

Families are classified as having traveled and

* They have children under 10 years of age
* They participated in a previous census in the same community
* They left the community for at least 8 weeks (2 months) for an area that has not received MDA in the past year and at least one child has returned and
* They have returned to reside in the community for at least 2 months

Sentinel Children: In all 52 communities, samples of 135 children will be selected from the community census lists every six months for survey and examination.

These children:

* must be between 1 year and 9.9 years of age,
* must be a resident in the community and not a short-term (less than 2 months) visitor,
* must not have an ocular condition that would preclude grading trachoma or taking an ocular specimen,
* must be willing to have a swab taken as part of being a sentinel child (this is critical, as each swab result counts towards the criteria for stopping MDA), and
* must have an identifiable guardian capable of providing consent to participate.

Adult Women: In all 52 communities, samples of 100 women will be selected from the baseline community census list.

These women:

* must be aged 15 years and over
* must be a resident in the community and not a short term (less than 2 months) visitor
* must not have an ocular condition that precludes grading of scarring on upper conjunctiva
* must be able to provide informed consent.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila K West, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] West SK, Munoz B, Mkocha H, Dize L, Gaydos CA, Swenor B, Ervin AM, Quinn TC. Treating village newcomers and travelers for trachoma: Results from ASANTE cluster randomized trial. PLoS One. 2017 Jun 29;12(6):e0178595. doi: 10.1371/journal.pone.0178595. eCollection 2017. PMID 28662043

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial was conducted at the community level and not at the participant level.Therefore, we are presenting the data only at the community level.
Units Other Than Participants: community
Groups:
- Intervention: Communities will receive usual care,including annual mass drug administration with azithromycin if trachoma infection level is greater than 1% or Follicular Trachoma (TF) is 5% or more. Communities will have MDA stopped if infection is 1% or less, or TF is less than 5%. MDA will be reinstated if infection re-emerges to 6% or more. In addition, surveillance and treatment with azithromycin of newcomer and traveler families within 2 weeks of arrival to or return to the community.
  Surveillance and treatment with azithromycin of newcomer and traveler families: The intervention is a surveillance for newcomers and travelers in communities, and provision of azithromycin to them at the time of arrival, in advance of scheduled mass drug administration
  Usual care: Scheduled MDA of azithromycin if trachoma infection level is greater than 1% or TF is 5% or more. Communities will have MDA stopped if infection is 1% or less, or TF is less than 5%. MDA will be reinstated if infection re-e
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | NA; 26 community (26 communities were randomized to intervention group The study was conducted at the community level.) | NA; 26 community (26 communities were randomized to control group The study was conducted at the community level.)
Completed | NA; 26 community (The study was conducted at the community level.) | NA; 26 community (The study was conducted at the community level.)
Not Completed | NA; 0 community | NA; 0 community

BASELINE CHARACTERISTICS:
Population: We collected and analyzed data on community level. Age and sex were not part of final analysis.
Units Other Than Participants: community
Groups:
- Intervention: Communities will receive usual care,including annual mass drug administration with azithromycin if trachoma infection level is greater than 1% or TF is 5% or more. Communities will have MDA stopped if infection is 1% or less, or TF is less than 5%. MDA will be reinstated if infection re-emerges to 6% or more. In addition, surveillance and treatment with azithromycin of newcomer and traveler families within 2 weeks of arrival to or return to the community.
  Surveillance and treatment with azithromycin of newcomer and traveler families: The intervention is a surveillance for newcomers and travelers in communities, and provision of azithromycin to them at the time of arrival, in advance of scheduled mass drug administration
  Usual care: Scheduled mass drug administration (MDA) of azithromycin if trachoma infection level is greater than 1% or TF is 5% or more. Communities will have MDA stopped if infection is 1% or less, or TF is less than 5%. MDA will be reinstated if infection re-e
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 26 | 26 | 52
Number analyzed (community) | 26 | 26 | 52
Age, Customized [Count of Units; unit: community]
  Age not analyzed at community level | NA — We collected and analyzed data on community level.Age was not part of final analysis. | NA — We collected and analyzed data on community level.Age was not part of final analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Units; unit: community] — We collected and analyzed data on community level.Sex was not part of final analysis.
  community
    Female | NA — We collected and analyzed data on community level.Sex was not part of final analysis. | NA — We collected and analyzed data on community level.Sex was not part of final analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — We collected and analyzed data on community level.Sex was not part of final analysis. | NA — We collected and analyzed data on community level.Sex was not part of final analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: community]
  Tanzania | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Communities With C. Trachomatis Infection Prevalence of 1% or Below
Description: The proportion of communities with C. trachomatis infection prevalence at 1% or below in children ages 1 to 9 years at the 24-month survey, comparing the intervention arm to the usual practice arm
Time Frame: 24 months
Population: The trial was conducted at the community level
Measure: Count of Units; unit: community
Units Other Than Participants: community
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | NA | NA
Number analyzed (community) | 26 | 26
community | 7 | 4
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p > 0.05, Regression, Logistic; Odds Ratio (OR) = 2.6, 95% CI 2-sided [0.56 to 11.9]; The null hypothesis was that we could further decrease infection to 1% or less in more of the communities in the surveillance intervention arm, compared to control communities

2. Secondary Outcome: The Proportion of Communities With Clinical Trachoma Prevalence of 5% or Below
Time Frame: 24 months
Population: The trial was conducted at the community level
Measure: Count of Units; unit: community
Units Other Than Participants: community
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | NA | NA
Number analyzed (community) | 26 | 26
community | 21 | 20
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 1, Fisher Exact; Mean Difference (Final Values) = 3.9

3. Secondary Outcome: The Mean of the Prevalence of Active Trachoma (TF) in Communities in Both Arms.
Description: Model the risk of active trachoma in intervention and control communities. We used the mean % and 95 % confidence interval as they present for a variable to describe the center of the population the sample represents and the precision of the estimate of that center.
  If the variable is normally distributed in the population, the probability is 95% that the true mean falls in the 95% confidence interval.
Time Frame: Baseline only
Population: The trial was conducted at the community level
Measure: Mean (95% Confidence Interval); unit: community
Units Other Than Participants: community
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | NA | NA
Number analyzed (community) | 26 | 26
community | 5.2 [3.7 to 6.6] | 4.9 [3.2 to 6.5]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 24 months. The Community Health Workers collected data on adverse events after each newcomer and traveler family was identified and treated.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No